CLINICAL TRIAL: NCT00230568
Title: A 12-Week, Multicenter, Open-Label Study to Evaluate the Effectiveness and Safety of Donepezil Hydrochloride (Aricept) in Hispanic Patients With Mild to Moderate Alzheimer's Disease
Brief Title: EARTH 413: A Study of Aricept in Hispanic Patients With Mild to Moderate Alzheimer's Disease (AD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: James Prodafikas, Study Director, Eisai Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2020-A001-413
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Alzheimer's Disease
Keywords: Mild to Moderate Alzheimer's Disease; Hispanic; Latino; Spanish-speaking
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

INTERVENTIONS:
Drug: Aricept

SUMMARY:
12-week, open-label study to evaluate the effectiveness and safety of donepezil hydrochloride in Hispanic patients with mild to moderate Alzheimer's Disease (AD) in the U.S.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients who self-identify as Hispanic and currently live in the United States.
* Age range: Patients >= 50 years.
* Sex distribution: both men and women. Women must be two (2) years post-menopausal or surgically sterile.
* MMSE scores between 10 and 26 (inclusive).
* Patients must have diagnostic evidence of AD (DSM-IV and NINCDS/ADRDA criteria) either prior to or at the screening visit. Patients with AD who may also have cerebrovascular disease as evidenced by risk factors such as hypertension, diabetes, elevated cholesterol levels, and smoking are also eligible to enroll in the study. In order to be enrolled, such patients' clinical conditions must be controlled, and it must be the investigator's opinion that the patient's primary diagnosis is AD, not vascular dementia. The diagnosis of AD must be recorded in the patient's clinical record prior to the baseline visit.
* CT or MRI within the last 12 months consistent with a diagnosis of AD without any other clinically significant comorbid pathologies found. Patients with vascular changes may be included provided that they do not meet NINDS-AIREN criteria for probable Vascular Dementia (VaD). A copy of the report will be required and should be appended to the case report form. If there has been a significant change in clinical status suggestive of stroke or other neurological disease in addition to AD with onset between the time of the last CT or MRI and the screening evaluation, the scan should be repeated during screening.
* All patients must be naïve to Aricept® treatment. Previous use of an approved or unapproved cholinesterase inhibitor (Exelon® , Cognex®, Reminyl®/Razadyne®, metrifonate, physostigmine) or memantine is allowed provided that the medication was discontinued at least 3 months prior to screening and that the discontinuation was not done for the purpose of enrolling the patient in this trial.
* Patients must reside in the community. (Residence in an assisted living facility is allowed.)
* Patients must have a reliable caregiver or family member who agrees to accompany the patient to all clinic visits, provide information about the patient as required by the protocol, and ensure compliance with the medication schedule. The caregiver must have a minimum of three days per week of direct contact with the patient (for at least 4 hours per day during waking hours).
* The patient must be capable of reliably completing study assessments including all efficacy parameters (MMSE, SDMT, and FOME) and all procedures scheduled during the screening, baseline and all follow-up visits.
* Patients must have clinical laboratory values within normal limits, and within the Eisai (sponsor) guidelines, or abnormalities considered not clinically significant by the investigator and sponsor.
* Patients with stable insulin-dependent diabetes or diabetes stabilized by diet and/or oral hypoglycemic agents are eligible provided they are monitored regularly to ensure adequacy of control. Patients with known diabetes should have an HbA1c of < 8% at screening.
* Patients with controlled hypertension (sitting diastolic BP < 95 mmHg), right bundle branch block (complete or partial), and pacemakers may be included in the study.
* Patients with thyroid disease also may be included in the study provided they are euthyroid and stable on treatment for at least 3 months prior to screening, and the stable treatment is maintained throughout study.
* Patients with a history of seizure disorder are allowed provided that they are on stable treatment for at least 3 months and have not had a seizure within the past 6 months.
* Patients must be able to swallow tablet medication -- no crushing of the tablet is allowed.
* Patient must be ambulatory or ambulatory-aided (i.e., walker or cane, or wheelchair). His/her vision and hearing (eyeglasses and/or hearing aid permissible) must be sufficient for compliance with testing procedures.

EXCLUSION CRITERIA:

* Age range: Patients < 50 years.
* MMSE score of < 10 or > 26.
* Patients with active or clinically significant conditions affecting absorption, distribution or metabolism of the study medication (e.g., inflammatory bowel disease, gastric or duodenal ulcers or severe lactose intolerance).
* Patients with a known hypersensitivity to piperidine derivatives or cholinesterase inhibitors.
* Patients without a reliable caregiver, or patients or caregivers who are unwilling or unable to complete any of the outcome measures and fulfill the requirements of this study.
* Patients who live in a skilled nursing facility (nursing home) or expect to enter nursing home within the next 3 months.
* Patients with clinically significant obstructive pulmonary disease or asthma not controlled with treatment at any time during the previous 3 months.
* Patients with recent (< 2 years) hematological/oncological disorders.
* Evidence of clinically significant, active gastrointestinal, renal, hepatic, endocrine or cardiovascular system disease.
* Patients with a current DSM-lV diagnosis of Major Depressive Disorder (MDD) or any current primary psychiatric diagnosis other than AD (as per DSM-lV).
* Patients with dementia complicated by delirium (DSM 290.30 or 290.11); depression or delusions are common in AD, and patients with severe symptoms so pronounced that they warrant an alternative, concurrent diagnosis, are excluded.
* Patients with a known or suspected history of alcoholism or drug abuse (within the past 5 years).
* Patients with treated vitamin B-12 deficiency who have not been on a stable dose of medication for at least 3 months prior to the study screening visit and who do not have normal serum B-12 levels at screening.
* Patients with treated hypothyroidism that have not been on a stable dose of medication for 3 months prior to screening and who do not have normal serum T-4 and TSH at screening.
* Patients with diabetes mellitus controlled by diet, oral medication, or insulin who do not have an HbA1c of < 8.0% and a random serum glucose value of < 170 mg/dl.
* Patients previously treated with Aricept® (donepezil Hydrochloride).
* Any condition which would make the patient or the caregiver, in the opinion of the investigator, unsuitable for the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-12; Primary Completion 2007-04 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
FOME (Fuld Object Memory Evaluation); SDMT (Symbol Digit Modalities Test); NPI (Neuropsychiatric Inventory); MMSE (the Mini-Mental State Examination). | 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: James Prodafikas, Study Director — Eisai Inc.
Locations (35):
- United States (35):
  - 21st Century Neurology, Phoenix, Arizona
  - Alzheimer's Disease and Cognitive Disorders Clinic at Barrow Neurology Institute, Phoenix, Arizona
  - Pacific Sleep Medicine Services, Inc., El Centro, California
  - Pacific Sleep Medicine Services, Inc., Los Angeles, California
  - Pacific Sleep Medicine Services, Inc., San Diego, California
  - Parkinson's Disease Movement Disorders Center - Boca Raton, Boca Raton, Florida
  - Bradenton Research Center, Bradenton, Florida
  - MD Clinical, Hallandale, Florida
  - Eastern Research, Hialeah, Florida
  - Berma Research Group, Hialeah, Florida
  - Cuervo Research Group, Miami, Florida
  - Seth Hochman, MD, Miami, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Ocala Neurodiagnostic Center, Ocala, Florida
  - Memory Disorder Center, Pompano Beach, Florida
  - Liliana Montoya, MD, Port Charlotte, Florida
  - Roskamp Institute Memory Clinic, Tampa, Florida
  - Palm Beach Neurology, West Palm Beach, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - The Northwestern Alzheimer's Center, Chicago, Illinois
  - Rush Alzheimer's Disease Center, Chicago, Illinois
  - Lozano, Cosme, MD, Joliet, Illinois
  - University of Nevada School of Medicine,, Las Vegas, Nevada
  - ClinSearch Inc., Kenilworth, New Jersey
  - University of New Mexico School of Medicine, Department of Psychiatry, Albuquerque, New Mexico
  - New York University School of Medicine, Aging and Dementia Research Center, New York, New York
  - The Burke Rehabilitation Hospital, White Plains, New York
  - North Carolina Neuropsychiatry, PA, Charlotte, North Carolina
  - Clinical Research Associates, Inc., Oklahoma City, Oklahoma
  - Clinical Research Center, Jenkintown, Pennsylvania
  - The Penn Ralston Center, University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Mental Sciences Insitute, Houston, Texas
  - Christopher Ticknor, MD, San Antonio, Texas
  - University of Texas, Health Science Center-San Antonio, San Antonio, Texas